CLINICAL TRIAL: NCT00359710
Title: Identity, Ancestry and Genetics: Patients' Perspectives
Brief Title: Patients' Perspectives on Identity, Ancestry and Genetics
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060148; 06-HG-0148
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-02-23

CONDITIONS: Family History
Keywords: Multiracial Populations; Human Genetic Variation; Family History; Admixture; Physician-Patient Communication; Ancestry; Self-Identified Multiracial Adults; Interview

SUMMARY:
This study will collect the opinions, understandings and personal health care experiences of multiracial persons of African and European ancestry. Understanding multiracial patients' beliefs and experiences about their race, ethnicity, ancestral origin and the genetic components of diseases can provide important data for developing ways to communicate how human genetic variation is related to self-identified race and ethnicity. The study will:

* Investigate multiracial individuals' beliefs about biological and genetic differences based on race and ethnicity;
* Collect stories of identity, ancestry and clinical experiences of multiracial individuals with one parent of African ancestry and one parent of European ancestry;
* Investigate multiracial patients' experiences regarding family health history and communication of genetic risk of disease.

Persons 21 years of age or older in the Atlanta, Georgia, or Washington, D.C., metropolitan areas who are from a multiracial background and have used health care services in the last 2 years may be eligible for this study. Participants are interviewed one-on-one for about 2 hours to gather information about their background, family ancestry, self-identity, race and ethnicity, health care interactions and genetics and health. Each participant completes a short questionnaire before and after the interview.

...

DETAILED DESCRIPTION:
The complex relationships between self-identified race, ethnicity, ancestral origin and the genetic components of diseases demands a better understanding of patients' conceptions of these identifiers and how they impact their health. The lived experiences of multiracial individuals can provide valuable perspectives on questions of race and ethnicity, the collection of ancestral information in assessing health history and communication of racial or ethnic specific disease risk. Understanding patients' beliefs and experiences will provide important data for developing ways to communicate how human genetic variation is related to self identified race and ethnicity. We aim to conduct semi-structured in-depth interviews with adults at least 21 years of age who identify as having a multiracial background with African and European ancestry. The study will include participants from the Atlanta, Georgia and Washington, D.C. metropolitan areas. This preliminary study uses qualitative methods to capture the personal stories of identity, ancestry and clinical experiences from a population that has not been adequately researched.

ELIGIBILITY:
* EXCLUSION CRITERIA:

Individuals will be excluded from the study if they do not have at least one parent that self-identifies as Black or has African ancestry and another parent that self identifies as White or has European ancestry. Other exclusion criteria include: (1) under 21 years of age, (2) not had at least two clinical visits with a health care professional in the last year and (3) not more than one individual per family.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-04-19; Study Completion 2011-02-23

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jorde LB, Wooding SP. Genetic variation, classification and 'race'. Nat Genet. 2004 Nov;36(11 Suppl):S28-33. doi: 10.1038/ng1435. PMID 15508000
- [Background] Collins FS. What we do and don't know about 'race', 'ethnicity', genetics and health at the dawn of the genome era. Nat Genet. 2004 Nov;36(11 Suppl):S13-5. doi: 10.1038/ng1436. PMID 15507997
- [Background] Bonham VL, Warshauer-Baker E, Collins FS. Race and ethnicity in the genome era: the complexity of the constructs. Am Psychol. 2005 Jan;60(1):9-15. doi: 10.1037/0003-066X.60.1.9. PMID 15641917